CLINICAL TRIAL: NCT01606202
Title: A Randomised, Double Blind, Placebo Controlled, Parallel Group Comparative Study of the Efficacy, Safety and Tolerability of Sublingual Cannabis Based Medicine Extracts and Placebo in Patients With Intractable Neuropathic Pain Associated With Spinal Cord Injury
Brief Title: A Study of Cannabis Based Medicine Extracts and Placebo in Patients With Pain Due to Spinal Cord Injury
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GWSC0101
Record Dates: First submitted 2012-05-21; First posted 2012-05-25 (Estimated); Results first posted 2012-09-28 (Estimated); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GW-1000-02 (Experimental): Active treatment.
  Interventions: Drug: GW-1000-02
- Placebo (Placebo Comparator): Placebo control.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GW-1000-02 — Contained delta-9-tetrahydrocannabinol (THC) (27 mg/ml):cannabidiol (CBD) (25 mg/ml) as extract of Cannabis sativa L., with peppermint oil, 0.05% (v/v), in ethanol:propylene glycol (50:50) excipient. Each actuation delivered 100 μl (THC 2.7 mg and CBD 2.5 mg). The maximum permitted dose of study medication was eight actuations in any three-hour period, and 48 actuations in any 24 hour period.
  Other Names: Sativex
  Arms: GW-1000-02
Drug: Placebo — Contained peppermint oil, 0.05% (v/v), quinoline yellow, 0.005% (w/v), sunset yellow, 0.0025% (w/v), in ethanol:propylene glycol (50:50) excipient. Each actuation delivered 100 μl. The maximum permitted dose of study medication was eight actuations in any three-hour period, and 48 actuations in any 24 hour period.
  Arms: Placebo

SUMMARY:
A study to investigate the effects of sublingual cannabis based medicine extracts on neuropathic pain associated with spinal cord injury.

DETAILED DESCRIPTION:
This was a multi-centre, double-blind, randomised, placebo-controlled, parallel-group study to evaluate the efficacy and tolerability of GW-1000-02 in central neuropathic pain associated with spinal cord injury. Patients were screened to determine eligibility and completed a seven to 21 day baseline period. Patients then returned to the centre for assessment, randomisation and initial dosing. Visits occurred at the end of treatment week one and at the end of the study (treatment week three) or upon withdrawal. Throughout the study, patients were permitted to take paracetamol as escape analgesic to relieve breakthrough pain. Patients in this study could elect to be screened for an open label extension study of GW-1000-02.

ELIGIBILITY:
Inclusion Criteria:

* Gave informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Diagnosis of non-acute spinal cord injury, with central neuropathic pain not wholly relieved by current therapy.
* Central neuropathic pain with a mean severity Numerical Rating Scale score at least four during last seven days of the baseline period.
* Relatively stable neurology during the preceding six months.
* Stable medication regimen during the preceding four weeks.
* Agreement, if female and of child bearing potential or if male with a partner of child bearing potential, to ensure that effective contraception was used during the study and for three months thereafter.
* Had not used cannabinoids for at least the preceding seven days and willing to abstain from any use of cannabinoids during the study.
* Clinically acceptable laboratory results at Visit 2.
* Ability (in the investigator's opinion) and willingness to comply with all study requirements.
* Agreement for the UK Home Office, their general practitioner, and their consultant if appropriate, to be notified of their participation in the study.

Exclusion Criteria:

* History of schizophrenia, other psychotic illness, severe personality disorder or other significant psychiatric disorder other than depression associated with their underlying condition.
* History of alcohol or substance abuse.
* Severe cardiovascular disorder, such as ischaemic heart disease, arrhythmias (other than well controlled atrial fibrillation), poorly controlled hypertension or severe heart failure.
* History of autonomic dysreflexia.
* History of epilepsy.
* If female, were pregnant or lactating, or were planning a pregnancy to occur during the course of the study.
* Significant renal or hepatic impairment.
* Elective surgery or other procedures requiring general anaesthesia scheduled to occur during the study.
* Terminal illness or were considered inappropriate for placebo medication.
* Any other significant disease or disorder which, in the opinion of the investigator, may have either put the subject at risk because of participation in the study, or may influenced the result of the study, or the subject's ability to participate in the study.
* Regular levodopa therapy within the seven days leading to study entry.
* If male, were receiving and were unwilling to stop sildenafil for the duration of the study.
* Known or suspected hypersensitivity to cannabinoids or any of the excipients of the study medications.
* Known or suspected adverse reaction to cannabinoids.
* Intention to travel internationally during the study.
* Intention to donate blood during the study.
* Participation in another research study in the 12 weeks leading to study entry.
* Previous randomisation into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2002-07; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal National Orthopaedic Hospital, Middlesex, United Kingdom

REFERENCES:
- [Derived] Thomas PA, Carter GT, Bombardier CH. A scoping review on the effect of cannabis on pain intensity in people with spinal cord injury. J Spinal Cord Med. 2022 Sep;45(5):656-667. doi: 10.1080/10790268.2020.1865709. Epub 2021 Jan 19. PMID 33465022

RESULTS

PARTICIPANT FLOW:
Groups:
- GW-1000-02: Each actuation of oromucosal spray delivers 2.7mg delta-9-tetrahydrocannabinol (THC) and 2.5mg cannabidiol (CBD). The maximum permitted dose of was eight actuations in any three hour period, and 48 actuations in any 24 hour period (THC 130 mg : CBD 120 mg).
- Placebo: Placebo control.The maximum permitted dose of was eight actuations in any three hour period, and 48 actuations in any 24 hour period.
Period: Overall Study
Arm/Group | GW-1000-02 | Placebo
Started | 56 | 60
Completed | 49 | 57
Not Completed | 7 | 3
Not completed — Adverse Event | 5 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Personal problems | 0 | 1
Not completed — Problems with administration | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GW-1000-02 | Placebo | Total
Number analyzed (Participants) | 56 | 60 | 116
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 51 | 55 | 106
  >=65 years | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (12.97) | 47.6 (12.69) | 48.1 (12.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 43 | 48 | 91
Region of Enrollment [Number; unit: participants]
  United Kingdom | 49 | 51 | 100
  Romania | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Central Neuropathic Pain 11-Point Numerical Rating Scale Scores at the End of Treatment (up to 51 Days).
Description: The Central Neuropathic Pain Numerical Rating Scale score was recorded three times daily, in the morning (on waking), at lunchtime and in the evening using the scale, 0 = 'No Pain' and 10 = 'Worst Possible Pain'. Patients were instructed to relate 'No Pain' to the time before the start of their spinal cord injury. End of Treatment was defined as the mean of the last seven days in the study or the mean of the last three days if the subject withdrew. A negative value indicates an improvement in pain score from baseline.
Time Frame: Up to 51 days
Population: All randomised patients who received at least one dose of test treatment and have on-treatment efficacy data were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- GW-1000-02: Contains THC (27 mg/ml) and CBD (25 mg/ml) delivered in 100 microlitre actuations by a pump action oromucosal spray. Maximum permitted dose was 48 actuations (THC 130 mg: CBD 120 mg) in 24 hours.
- Placebo: Contains no active drug but colourants and excipients. Maximum permitted dose was 48 actuations in 24 hours.
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 55 | 59
units on a scale | -0.74 (1.12) | -0.69 (1.39)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; The change in the pain Numerical Rating Scale score from baseline to End of Treatment was compared between treatment groups using analysis of covariance (ANCOVA). The model included treatment and centre as factors and baseline Numerical Rating Scale pain mean score as a covariate; Test type: Superiority or Other; p = 0.708, ANCOVA; Estimated mean treatment difference = -0.08, 95% CI 2-sided [-0.51 to 0.35]

2. Secondary Outcome: Change From Baseline in the Mean Percentage of Days on Which Escape Medication Was Used at the End of Treatment
Description: The percentage of days that subjects used escape medication was analysed and is presented as the mean change from baseline at the end of treatment. A negative value from baseline indicates an improvement.
Time Frame: Up to 51 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 55 | 59
percentage of days | -4.68 (18.25) | -2.91 (20.83)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; The change from baseline to End of Treatment in the percentage of days on which escape medication was used was compared between treatment groups using ANCOVA. The model included treatment and centre as factors and percentage of days on which escape medication was used as a covariate; Test type: Superiority or Other; p = 0.852, ANCOVA; Estimated mean treatment difference = -0.57, 95% CI 2-sided [-6.62 to 5.48]

3. Secondary Outcome: Change From Baseline in Mean Spasm Severity Numerical Rating Scale Score at the End of Treatment
Description: Each day, just before going to bed, patients recorded in their patient diary whether they experienced any spasms that day and, if yes, recorded the overall level of the spasm(s) experienced using an Numerical Rating Scale spasm scale ranging from 0 = "Mildest ever spasm" to 10 = "Worst ever spasm". The mean spasm severity scores were summarised and analysed analogously to the primary endpoint. A negative value from baseline indicates an improvement.
Time Frame: Up to 51 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 42 | 48
units on a scale | -0.50 (1.46) | -0.69 (1.59)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; The change from baseline to End of Treatment in the Spasm severity Numerical Rating Scale score was compared between treatment groups using ANCOVA. The model included treatment and centre as factors and the Spasm severity Numerical Rating Scale score as a covariate; Test type: Superiority or Other; p = 0.860, ANCOVA; Estimated mean treatment difference = 0.05, 95% CI 2-sided [-0.54 to 0.65]

4. Secondary Outcome: Change From Baseline in the Percentage of Days on Which Spasm Was Experienced at the End of Treatment
Description: Each day, just before going to bed, patients recorded in their patient diary whether they experienced any spasms that day. The percentage of days on which spasm was experienced were summarised and analysed analogously to the primary endpoint. A negative value from baseline indicates an improvement.
Time Frame: Up to 51 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 52 | 59
percentage of days | -1.92 (20.01) | -1.57 (22.62)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; The change from baseline to End of Treatment in the percentage of days on which spasm was experienced was compared between treatment groups using ANCOVA. The model included treatment and centre as factors and the Spasm percentage of days on which spasm was experienced as a covariate; Test type: Superiority or Other; p = 0.873, ANCOVA; Estimated mean treatment difference = -0.64, 95% CI 2-sided [-8.56 to 7.27]

5. Secondary Outcome: Change From Baseline in Mean Spasticity Severity Numerical Rating Scale Scores the End of Treatment.
Description: Each day at bed time patients recorded whether they experienced any spasticity that day and, if yes, the overall level of spasticity experienced was quantified using an Numerical Rating Scale from 0 = "Mildest ever spasticity" to 10 = "Worst ever spasticity". The mean spasticity severity scores and the changes from baseline to End of Treatment were to be calculated. A negative value indicates an improvement from baseline.
Time Frame: 0 - 51 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 35 | 43
units on a scale | -0.37 (1.25) | -0.46 (1.80)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; The change from baseline to End of Treatment in the spasticity severity Numerical Rating Scale score was compared between treatment groups using ANCOVA. The model included treatment and centre as factors and the baseline spasticity severity Numerical Rating Scale score as a covariate; Test type: Superiority or Other; p = 0.830, ANCOVA; Estimated mean treatment difference = 0.07, 95% CI 2-sided [-0.61 to 0.75]

6. Secondary Outcome: Change From Baseline in the Percentage of Days on Which Spasticity Was Experienced at the End of Treatment
Description: Each day, just before going to bed, patients recorded in their patient diary whether they had experienced any spasticity that day or not. The percentage of days on which spasticity was experienced (spasticity incidence) was calculated and summarised analogously to the primary efficacy parameter of Numerical Rating Scale pain score. A negative value from baseline indicates an improvement.
Time Frame: Up to 51 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 50 | 59
percentage of days | 0.86 (6.71) | 0.48 (14.76)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; The change from baseline to End of Treatment in the percentage of days on which spasticity was experienced was compared between treatment groups using ANCOVA. The model included treatment and centre as factors and the percentage of days on which spasticity was experienced as a covariate; Test type: Superiority or Other; p = 0.860, ANCOVA; Estimated mean treatment difference = 0.40, 95% CI 2-sided [-4.08 to 4.88]

7. Secondary Outcome: Change From Baseline in Modified Ashworth Scale Score at the End of Treatment
Description: The Modified Ashworth Scale is a five-point scale conducted on four pre-identified muscle groups. Only the lower limb was assessed because not all Spinal Cord Injury patients upper limb disability. The assessor used the Modified Ashworth scale ranging from 0 ("No increase in muscle tone") to 4 ("Affected part(s) rigid in flexion or extension") to rate the muscle tone for knee and ankle for the left and right sides separately at a pre-dose visit and at the end of treatment. The average of the four individual scores and was taken. A negative value indicates an improvement from baseline.
Time Frame: Up to 51 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 40 | 44
units on a scale | -0.13 (0.43) | -0.01 (0.42)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; The change from baseline to End of Treatment in the Modified Ashworth scale score was compared between treatment groups using ANCOVA. The model included treatment and centre as factors and the Modified Ashworth scale score as a covariate; Test type: Superiority or Other; p = 0.142, ANCOVA; Estimated mean treatment difference = -0.14, 95% CI 2-sided [-0.33 to 0.05]

8. Secondary Outcome: Change From Baseline in the Mean Short Orientation Memory Function Concentration Test Score at the End of Treatment
Description: Patients were asked at baseline and end of treatment, to complete the Short Orientation Memory Function Concentration Test as a measure of cognitive function. The minimum score is 0 and maximum of 28 which denoted good cognitive function .
  A negative value from baseline indicates a deterioration.
Time Frame: Up to 51 days
Population: All patients who were randomised, received at least one actuation of study medication and had on-treatment efficacy data were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 55 | 58
units on a scale | 0.4 (2.79) | 0.2 (2.98)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; The change from baseline in the mean Short Orientation Memory Concentration score, was compared between treatment groups using ANCOVA. The model included treatment and centre as factors and baseline Short Orientation Memory Concentration test score as a covariate; Test type: Superiority or Other; p = 0.824, ANCOVA; Estimated mean treatment difference = -0.11, 95% CI 2-sided [-1.13 to 0.90]

9. Secondary Outcome: Change From Baseline in Mean Spitzer Quality of Life Index Score at the End of Treatment
Description: The Spitzer Quality of Life Index questionnaire consists of five sections, relating to activity, daily living, health, support and outlook. Each section has three choices (numbered 1, 2 and 3) and the patient is required to choose the one that best describes their quality of life during the last week. Choice 1 is scored 2, choice 2 is scored 1 and choice 3 is scored 0. The total Spitzer is the unweighted sum of the five scores. The scale is 0 (bad) to 10 (good). A positive value indicates an improvement from baseline.
Time Frame: Up to 51 days
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 55 | 58
units on a scale | 0.1 (1.41) | 0.1 (1.30)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; The change from baseline to End of Treatment in the Spitzer Quality of Life Index score was compared between treatment groups using ANCOVA. The model included treatment and centre as factors and the Spitzer Quality of Life Index score as a covariate; Test type: Superiority or Other; p = 0.847, ANCOVA; Estimated mean treatment difference = -0.04, 95% CI 2-sided [-0.49 to 0.40]

10. Secondary Outcome: Change From Baseline in the Mean Caregiver Strain Index Score at the End of Treatment
Description: Carers were asked at baseline and end of treatment to complete the Caregiver Strain Index, as a measure of the strain they felt from being a carer, the maximum possible score being 13. A negative value from baseline indicates an improvement.
Time Frame: Up to 51 days
Population: All caregivers of patients in the current study who responded to the caregiver strain index questionnaire were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 12 | 16
units on a scale | -0.3 (2.73) | 1.2 (3.45)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; The change from baseline to End of Treatment in the Caregiver Strain Index score was compared between treatment groups using ANCOVA. The model included treatment and centre as factors and the baseline Caregiver Strain Index score as a covariate; Test type: Superiority or Other; p = 0.287, ANCOVA; Estimated mean treatment difference = -1.29, 95% CI 2-sided [-3.74 to 1.16]

11. Secondary Outcome: Number of Subjects Who Reported an Improvement in Their Overall Condition in the Patient Global Impression of Change at the End of Treatment
Description: The Patient Global Impression of Change asked patients to give their impression of the overall change in their condition during the study at the end of treatment using the following scale: 1 = Very Much Improved, 2 = Much Improved, 3 = Minimally Improved, 4 = No Change, 5 = Minimally Worse, 6 = Much Worse, 7 = Very Much Worse. The number of patients who scored their condition as 1, 2, or 3 (improved) is presented.
Time Frame: Up to 51 days
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 56 | 60
participants | 30 | 12
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; The proportion of subjects who considered their condition 'Very Much Improved', 'Much Improved' or 'Minimally Improved' was compared between treatment groups using Fisher's Exact Test; Test type: Superiority or Other; p < 0.001, Fisher Exact; Estimated mean treatment difference = 33.86, 95% CI 2-sided [17.07 to 50.64]

12. Secondary Outcome: Change From Baseline in the Mean Brief Pain Inventory Score at the End of Treatment
Description: The Brief Pain Inventory is a 14-item questionnaire that asks patients to rate pain over the prior week and the degree to which it interferes with activities on a 0 to 10 scale, where 0=no pain and 10=pain as bad as you can imagine. Severity is measured as worst pain, least pain, average pain, and pain right now. The severity composite score is calculated as the arithmetic mean of the four severity items(range 0-10). A negative value indicates an improvement in worst pain score from baseline.
Time Frame: 0 - 51 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 53 | 57
units on a scale | -3.1 (5.22) | -1.2 (4.64)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; The change from baseline to End of Treatment in the Brief Pain Inventory score was compared between treatment groups using ANCOVA. The model included treatment and centre as factors and baseline Brief Pain Inventory score as a covariate; Test type: Superiority or Other; p = 0.032, ANCOVA; Estimated mean treatment difference = -1.93, 95% CI 2-sided [-3.69 to -0.16]

13. Secondary Outcome: Change From Baseline in the Mean Sleep Disturbance Numerical Rating Scale Score at the End of Treatment
Description: Each day patients recorded in their patient diary whether they woke during the previous night using the following scoring system: 0 = No, 1 = Once, 2 = Twice, 3 = More than twice, 4 = Awake most of the night. A negative value indicates an improvement from baseline.
Time Frame: 0 - 51 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 55 | 59
units on a scale | -0.41 (0.59) | -0.38 (0.73)

14. Secondary Outcome: Incidence of Adverse Events as a Measure of Patient Safety.
Description: The number of patients who experienced an adverse event during the study is presented.
Time Frame: Up to 61 days
Population: All randomised patients who received at least one dose of study drug were included in the Safety population.
Measure: Number; unit: participants
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 56 | 60
participants | 46 | 29

ADVERSE EVENTS:
Time Frame: All adverse events occurring from the time of consent to post study follow up (0-61 days) were collected. All deaths and serious adverse events occurring within 28 days of the final dose of study medication were also collected.
Description: All adverse events occurring during the study were reported on the running logs at the back of the study case report form.
Arm/Group | GW-1000-02 | Placebo
Serious Adverse Events (participants affected / at risk) | 3/56 | 2/60
Other Adverse Events (participants affected / at risk) | 46/56 | 29/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GW-1000-02 (N=56) | Placebo (N=60)
Anaemia Not Otherwise Specified Aggravated (Blood and lymphatic system disorders) | 1 | 0
Fall (General disorders) | 1 | 1
Methicillin-resistant Staphylococcus aureus infection (Infections and infestations) | 1 | 0
Bladder Infection Not Otherwise Specified (Infections and infestations) | 0 | 1
Pneumonia Not Otherwise Specified (Infections and infestations) | 0 | 1
Tibia Fracture (Injury, poisoning and procedural complications) | 1 | 0
Upper Limb Fracture Not Otherwise Specified (Injury, poisoning and procedural complications) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Confusion (Psychiatric disorders) | 1 | 0
Paranoia (Psychiatric disorders) | 1 | 0
Contusion (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GW-1000-02 (N=56) | Placebo (N=60)
Nausea (Gastrointestinal disorders) | 6 | 3
Constipation (Gastrointestinal disorders) | 4 | 0
Dry Mouth (Gastrointestinal disorders) | 4 | 0
Oral Pain (Gastrointestinal disorders) | 2 | 3
Lethargy (General disorders) | 4 | 0
Feeling Abnormal (General disorders) | 3 | 0
Feeling Drunk (General disorders) | 3 | 0
Urinary Tract Infection Not Otherwise Specified (Infections and infestations) | 8 | 4
Alanine Aminotransferase Increased (Investigations) | 2 | 3
Gamma-Glutamyltransferase Increased (Investigations) | 2 | 3
Dizziness (Nervous system disorders) | 14 | 5
Dysgeusia (Nervous system disorders) | 9 | 4
Somnolence (Nervous system disorders) | 7 | 0
Headache Not Otherwise Specified (Nervous system disorders) | 5 | 0
Disturbance in Attention (Nervous system disorders) | 3 | 0
Vision Blurred (Eye disorders) | 2 | 0
Oral Discomfort (Gastrointestinal disorders) | 2 | 0
Vomiting Not Otherwise Specified (Gastrointestinal disorders) | 2 | 0
Application Site Pain (General disorders) | 2 | 0
Fatigue (General disorders) | 2 | 0
Pain Exacerbated (General disorders) | 2 | 0
Fall (General disorders) | 0 | 2
Feeling of Relaxation (General disorders) | 0 | 2
Pyrexia (General disorders) | 0 | 2
Blood Bilirubin Increased (Investigations) | 2 | 0
Blood Sodium Decreased (Investigations) | 2 | 0
Haematocrit Decreased (Investigations) | 2 | 0
Haemoglobin Decreased (Investigations) | 2 | 0
Red Blood Cell Count Decreased (Investigations) | 2 | 0
White Blood Cell Count Increased (Investigations) | 2 | 0
Neutrophil Count Increased (Investigations) | 0 | 2
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 2
Speech Disorder (Nervous system disorders) | 2 | 0
Paraesthesia (Nervous system disorders) | 0 | 2
Confusion (Psychiatric disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 2
Flushing (Vascular disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GW will coordinate the dissemination of data from this study and may solicit input and assistance from the principal investigator. All publications, for example manuscripts, abstracts, oral/slide presentations or book chapters based on this study, must be submitted to GW for corporate review before release.